CLINICAL TRIAL: NCT05816434
Title: Can More Sleep Improve Pain Responses, Symptomatology, and Regulation in College Students?
Brief Title: More Sleep: Pain Response to Longer Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Anne-Marie Chang, Associate Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00022196
Record Dates: First submitted 2023-03-20; First posted 2023-04-18 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Sleep; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Extension (Experimental): 1 week of >1 hour increased time in bed
  Interventions: Behavioral: Sleep extension
- Control (No Intervention): Sustained sleep behavior

INTERVENTIONS:
Behavioral: Sleep extension — >1 hour additional time in bed per night for 1 week.
  Arms: Sleep Extension

SUMMARY:
This study is being done to find out whether extending sleep for at least an hour per night, seven days a week, predicts a higher tolerance and a higher threshold for pain. This is a 21-day study. Participants will be asked to wear sleep- and heart- monitoring watches. Pressure pain and cold pain will be measured at study visits.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 24 (inclusive) years of age at enrollment
2. Fluent English speaker and reader
3. Willing to refrain from initiating new therapeutic interventions (e.g., medication; behavioral) designed to target sleep or pain for the duration of study participation

Exclusion Criteria:

1. Diagnosed with a sleep disorder
2. Diagnosed with a pain disorder
3. Has experienced a cold-related injury frostbite or has any other nerve damage to the feet
4. Has a history of injury to any of the muscular measurement sites for pain (I.e. shoulder, jaw, forearm)
5. Diagnosed with hypertension or cardiovascular disease
6. Evidence of hypertension
7. Diagnosed serious mental health disorder or substance use disorder
8. Taking any physician-directed pharmacologic intervention for sleep
9. Taking any physician-directed pharmacologic intervention for pain
10. Personal health history of traumatic brain injury
11. Pregnant
12. Current smoker

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-11-04 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Change in pressure pain threshold from before to after sleep extension | Momentary at study visit 2 (at the end of week1) and a week later at study visit 3 (at the end of week2).
  Bilateral response to a clinically standard algometer at 3 different physical palpation sites. A higher pressure reading indicates a better pain response.
Change in pressure pain tolerance from before to after sleep extension | Momentary at study visit 2 (at the end of week1) and a week later at study visit 3 (at the end of week2).
  Bilateral response to a clinically standard algometer at 3 different physical palpation sites. A higher pressure reading indicates a better pain response.
Change in weekly average of momentary pain self-reports from before to after sleep extension | (averaged) Daily surveys during study week 1 (pre-intervention) and study week 2 (intervention)
  Intermittent pain intensity using a Visual Analog Scale (0-100, where 0 = "no pain", 100 = "worst pain imaginable in current circumstances"). Higher values indicated more pain, and a negative change indicates a decrease in pain.
Change in thermal pain threshold from before to after sleep extension | Momentary at study visit 2 (at the end of week1) and a week later at study visit 3 (at the end of week2).
  Latency to respond to a bilateral cold pressor test (feet). A longer latency to threshold indicates better pain response.
Change in thermal pain tolerance from before to after sleep extension | Momentary at study visit 2 (at the end of week1) and a week later at study visit 3 (at the end of week2).
  Latency to respond to a bilateral cold pressor test (feet). A longer latency to tolerance indicates better pain response.
Change in pain inhibition from before to after sleep extension | Momentary at study visit 2 (at the end of week1) and a week later at study visit 3 (at the end of week2).
  Pain inhibition is measured as the difference in pressure pain threshold from before to after cold pressor procedure. A reduction in pressure pain threshold is typical after cold pressor procedure. A greater reduction in pain threshold indicates a better response of the pain inhibitory system.

CONTACTS AND LOCATIONS:
Locations (1):
- Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Time Frame: The data will be shared within one year after the first publication related to primary outcomes.
Access Criteria: Request for data should be made in writing to the PI.